CLINICAL TRIAL: NCT00192491
Title: A Randomized, Placebo-Controlled, Trial to Assess Safety, Tolerability, and Immunogenicity of Influenza Virus Vaccine, Trivalent, Types A & B, Live Cold-Adapted (FluMist) and Measles, Mumps, Rubella, (MMRIIÒ) and Varicella (VARIVAXÒ) Vaccines Administered Concurrently to Healthy Children (AV018)
Brief Title: Trial to Assess Safety, Tolerability, and Immunogenicity of Influenza Virus Vaccine, Trivalent, Types A & B, Live Cold-Adapted (FluMist) and Measles, Mumps, Rubella, and Varicella Vaccines Administered Concurrently to Healthy Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Robert Walker, M.D., MedImmune Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: AV018
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2008-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 (Active Comparator): FluMist
  Interventions: Biological: FluMist
- 3 (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- 1 (Active Comparator): FluMist with other solution
  Interventions: Biological: FluMist

INTERVENTIONS:
Biological: FluMist — Nasal Sprayer of one dosage of FluMist and other experimental
  Arms: 1
Biological: FluMist — Nasal sprayer of FluMist
  Arms: 2
Other: Placebo — Nasal Sprayer of Placebo
  Arms: 3

SUMMARY:
* To compare immune responses to measles, mumps, rubella, and varicella antigens following vaccination in children who receive FluMist concurrently with MMRIIÒ and VARIVAXÒ and in children who receive an intranasal placebo mist concurrently with MMRIIÒ and VARIVAXÒ (Group 2 vs. Group 1).
* To compare immune responses to the three strains of influenza (H1N1, H3N2, and B) following a two dose regimen of FluMist in children who receive the initial FluMist dose concurrently with MMRIIÒ and VARIVAXÒ and in children who receive two doses of FluMist alone (Group 2 vs. Group 3).Secondary:
* To assess the safety and tolerability of concurrent administration of FluMist with MMRIIÒ and VARIVAXÒ.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 15 months of age (not reached their 16th month birthday);
* In good health;
* Parent/guardian available by telephone or for home visits;
* Ability of the parent/guardian to understand and comply with the requirements of the protocol;
* Signed informed consent by parent/guardian; and
* Up to date with the primary series of recommended vaccines per standard clinic practice and local vaccine availability.

Exclusion Criteria:

* Previous known measles, mumps, rubella or varicella disease;
* Previous vaccination against measles, mumps, rubella or varicella disease;
* Hypersensitivity to egg or egg protein;
* Signs or symptoms of any immunosuppressive or immune deficiency disease or ongoing immunosuppressive therapy; or an immunosuppressed individual living in the same household;
* Acute febrile (>100.0oF [37.8°C] oral) illness or clinically significant upper respiratory illness within the 72 hours prior to enrollment;
* Use of aspirin (acetylsalicylic acid) or aspirin-containing products in the month prior to enrollment, or expected use of aspirin while enrolled in this study;
* Administration of any intranasal medication within two weeks prior to enrollment or expected receipt during this study;
* Administration of any live virus vaccine within one month prior to enrollment through 30 days after Visit 3;
* Administration of any inactivated vaccine within two weeks prior to enrollment through 30 days after Visit 3;
* Participation in another investigational trial within one month prior to enrollment or expected enrollment in another investigational trial during this study;
* Receipt of any blood product within three months prior to vaccination or expected receipt within the study duration; and
* Any condition which, in the opinion of the investigator, would interfere with the interpretation or evaluation of the vaccines.
* History of two or more episodes of medically attended wheezing illness by parent/guardian report.
* History of medically attended wheezing illness or bronchodilator medication use within four weeks of enrollment by parent/guardian report.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2000-12; Primary Completion 2003-09 (Estimated); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
compare immune responses to measles, mumps, rubella, and varicella antigens following vaccination in children who receive FluMist concurrently with MMRIIÒ and VARIVAXÒ and in children | Day 42

SECONDARY OUTCOMES:
Compare immune responses to the three strains of influenza (H1N1, H3N2, and B) following a two dose regimen of FluMist in children who receive the initial FluMist | Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, M.D., Study Director — MedImmune LLC

REFERENCES:
- [Derived] Nolan T, Bernstein DI, Block SL, Hilty M, Keyserling HL, Marchant C, Marshall H, Richmond P, Yogev R, Cordova J, Cho I, Mendelman PM; LAIV Study Group. Safety and immunogenicity of concurrent administration of live attenuated influenza vaccine with measles-mumps-rubella and varicella vaccines to infants 12 to 15 months of age. Pediatrics. 2008 Mar;121(3):508-16. doi: 10.1542/peds.2007-1064. PMID 18310199